CLINICAL TRIAL: NCT05955755
Title: The Effect of Butterfly Vacuum Blood Collection Set and Standard Vacutanier Needle Used in Blood Collection in Children on the Level of Pain and Fear: A Randomized Controlled Study
Brief Title: The Effect of Butterfly Vacuum Blood Collection Set and Standard Vacutanier Needle on the Level of Pain and Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Özlem Selime MERTER, ASSISTANT PROFESSOR, Firat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023/ 08- 10
Record Dates: First submitted 2023-07-11; First posted 2023-07-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Child Development; Nursing Caries; Pain; Fear
Keywords: child; nurse; fear; pain; blood collection
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): A butterfly vacuum blood collection set will be used in the blood collection process from the children in the experimental group.
  Interventions: Other: butterfly vacuum blood collection set
- control group (No Intervention): A standard vacutanier needle will be used for blood collection from the children in the control group. Vacutanier needle is used routinely in the blood collection unit where the study will be performed.

INTERVENTIONS:
Other: butterfly vacuum blood collection set — Blood collection from the children in the experimental group will be performed with a butterfly vacuum blood collection set.
  Arms: experimental group

SUMMARY:
This study was planned to examine the effects of the butterfly vacuum blood collection set and standard vacutanier needle used during blood collection in children on the level of pain and fear. It is a randomized controlled trial.The study will be conducted in the pediatric blood collection unit with children between the ages of 7 and 12 who have undergone blood tests by a pediatrician.Data collection tools: "Descriptive Information Form", "Difficult Intravenous Intervention Score" for Children, "Numerical Pain Scale", "Child Fear Scale" will be used to collect data.The data will be uploaded to the computer and coded by the researchers, and the data will be evaluated in the SPSS package program. The sociodemographic data of the children participating in the study will be given as numbers and percentage distributions. Appropriate tests will be used by analyzing the data for normal distribution. The statistical significance level of the study was determined as p< 0.05. In addition, at the end of the research, the status of working with sufficient sample size will be tested with post-hoc power analysis.

DETAILED DESCRIPTION:
Purpose of the study: This study was planned to examine the effects of the butterfly vacuum blood collection set and standard vacutanier needle used during blood collection in children on the level of pain and fear.

Type of Study: It is a randomized controlled study. Location and Characteristics of the Study: It will be conducted in the pediatric blood collection unit of Fırat University Hospital, with children aged 7-12 who are subjected to blood tests by a pediatrician.

Population-Sample: The population of the study will consist of children who applied for blood collection in the pediatric blood collection unit of Fırat University Hospital. A pilot study will be conducted to determine the number of samples. For the pilot study, 20 participants will be taken from each group and a total of 40 samples will be taken. As a result of the pilot study, power analysis will be performed and the number of samples will be determined. Randomization will be done to assign the participants to the groups. Grouping will be done using simple random sampling. Randomization will be provided using the Random Sequence Generator on the www.random.org website. Each participant who volunteers to participate in the study and meets the criteria will be given a number. Accordingly, which number will take place in which group will be determined in advance.

Data collection tools: "Descriptive Information Form", "Difficult Intravenous Intervention Score" for Children, "Numerical Pain Scale", "Child Fear Scale" will be used to collect data.

Data Collection: Data collection Children who accept to participate in the 1st stage study will be given the Difficult Intravenous Intervention Score for Children.

In the 2nd stage, an Introductory Information Form and Child Fear Scale will be used for children whose Difficulty Intravenous Intervention Score for Children is below 4.

In the 3rd phase, children who meet the research criteria will be randomized. In stage 4, blood collection from children will be performed by the same nurse (a volunteer nurse with 5 years of experience in pediatric phlebotomy). A butterfly vacuum blood collection set will be used for blood collection from the children in the experimental group, and a standard vacutanier needle will be used for the blood collection from the children in the control group.

In the 5th stage, children will be evaluated for pain and fear after bloodletting. This assessment will be made by the child, parent and nurse.

Evaluation of the data: The data will be uploaded to the computer and coded by the researchers, and the data will be evaluated in the SPSS package program. The sociodemographic data of the children participating in the study will be given as numbers and percentage distributions. Appropriate tests will be used by analyzing the data for normal distribution. The statistical significance level of the study was determined as p< 0.05. In addition, at the end of the research, the status of working with sufficient sample size will be tested with post-hoc power analysis.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 7-12

  * Do not have a chronic disease
  * Peripheral intravenous catheter (PIC) application by the same nurse (with at least 5 years of experience)
  * Able to express oneself verbally
  * No visual and auditory problems
  * Forced intravenous access score below 4

Exclusion Criteria:

* Children treated with tropical anesthetic before the procedure

  * Children who have taken analgesics in the last 6 hours
  * Neurodevelopmentally delayed children
  * Children with chronic disease
  * Children with unsuccessful blood draw attempts

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-09-24 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Scale | 1 day
  This method, which is aimed at determining the severity of pain, aims to explain the patient's pain in numbers. Absence of pain (0) is evaluated as unbearable pain (10) on numerical scales.

OTHER OUTCOMES:
Challenging Intravenous Intervention Score for Children | 1 day
  Visibility of the vein is scored as visible = 0, invisible = 2 points. The palpability of the vein is scored as palpable = 0, non-palpable = 2 points. Age status is scored as ≥ 36 months = 0, 12-35 months = 1, < 12 months = 3 points. In the variable of prematurity, children with a gestational age before 38 weeks are considered premature and scored as not premature = 0, premature = 3 points. The skin tone variable is evaluated as light and dark, scored as light = 0 and dark = 1. Skin tone cards of Dermablend cosmetics company were used for the skin tone variable (numbers 11 from light to dark skin, numbers 1-2-4-5 fair skin, numbers 3-6-7-8-9-10-11 dark skin). The score that can be obtained from this score varies between 0-11, if the score obtained from the score is four or more, the vascular access is considered difficult with a 50% probability of failure.
Child Fear Scale | 1 day
  This Scale includes 5 different facial expressions. This scale is scored between 0 and 4, and it is stated to be a reliable and valid measurement tool in the evaluation of fear.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Karaarslan, Study Chair — Manisa Celal Bayar University; Atiye Karakul, Study Chair — Tarsus University
Locations (1):
- Fırat Univesity, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKinley S, Coote K, Stein-Parbury J. Development and testing of a Faces Scale for the assessment of anxiety in critically ill patients. J Adv Nurs. 2003 Jan;41(1):73-9. doi: 10.1046/j.1365-2648.2003.02508.x. PMID 12519290
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] O'Conner-Von S. Preparing children for surgery--an integrative research review. AORN J. 2000 Feb;71(2):334-43. doi: 10.1016/s0001-2092(06)62113-3. PMID 10707264
- [Background] Thompson RH, Vernon DT. Research on children's behavior after hospitalization: a review and synthesis. J Dev Behav Pediatr. 1993 Feb;14(1):28-35. PMID 8432876
- [Background] Yen K, Riegert A, Gorelick MH. Derivation of the DIVA score: a clinical prediction rule for the identification of children with difficult intravenous access. Pediatr Emerg Care. 2008 Mar;24(3):143-7. doi: 10.1097/PEC.0b013e3181666f32. PMID 18347490
- [Background] Inal S, Kelleci M. The Effect of External Thermomechanical Stimulation and Distraction on Reducing Pain Experienced by Children During Blood Drawing. Pediatr Emerg Care. 2020 Feb;36(2):66-69. doi: 10.1097/PEC.0000000000001264. PMID 28885392
- [Background] Coventry LL, Jacob AM, Davies HT, Stoneman L, Keogh S, Jacob ER. Drawing blood from peripheral intravenous cannula compared with venepuncture: A systematic review and meta-analysis. J Adv Nurs. 2019 Nov;75(11):2313-2339. doi: 10.1111/jan.14078. Epub 2019 Jun 20. PMID 31115075
- [Background] Ozalp Gerceker G, Ayar D, Ozdemir EZ, Bektas M. Effects of virtual reality on pain, fear and anxiety during blood draw in children aged 5-12 years old: A randomised controlled study. J Clin Nurs. 2020 Apr;29(7-8):1151-1161. doi: 10.1111/jocn.15173. Epub 2020 Jan 22. PMID 31889358
- [Background] Celikol S, Tural Buyuk E, Yildizlar O. Children's Pain, Fear, and Anxiety During Invasive Procedures. Nurs Sci Q. 2019 Jul;32(3):226-232. doi: 10.1177/0894318419845391. PMID 31203776
- [Background] Sapci E, Bilsin Kocamaz E, Gungormus Z. Effects of applying external cold and vibration to children during vaccination on pain, fear and anxiety. Complement Ther Med. 2021 May;58:102688. doi: 10.1016/j.ctim.2021.102688. Epub 2021 Feb 26. PMID 33640458